CLINICAL TRIAL: NCT02527837
Title: The Effect of Sodium Nitrite Infusion on Renal Variables, Peripheral and Central Blood Pressure in Hypertensive Versus Normotensive Subjects in a Randomised, Placebo Controlled, Cross Over, Case-control Study
Brief Title: The Effect of Sodium Nitrite on Renal Function and Blood Pressure in Hypertensive Versus Healthy Subjects
Acronym: HYCA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, Chief physician, professor, DMSc, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: JBR-1-2014
Record Dates: First submitted 2015-02-18; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Sodium Nitrite; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium nitrite (Active Comparator): Sodium nitrite, 240 micrograms/kg/hour for 2 hours
  Interventions: Drug: Sodium nitrite
- Placebo (Placebo Comparator): Sodium chloride, isotonic 0.9%, 25 ml/hour for 2 hours
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Sodium nitrite — Sodium nitrite, 240 micrograms/kg/hour for 2 hours
  Other Names: NaNO2
  Arms: Sodium nitrite
Drug: Sodium chloride — Sodium chloride, isotonic 0.9%, 25 ml/hour for 2 hours
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate how the effect of infused sodium nitrite differs in hypertensives compared to healthy age and sex matched controls. The effects on renal handling of nitrite, nitrate, sodium and water, plasma concentrations of vasoactive hormones, peripheral (brachial) and central blood pressure will be evaluated.

DETAILED DESCRIPTION:
Nitric oxide (NO) is an important vasodilating molecule with a very complex biochemistry and metabolism. NO is classically synthesized from L-arginin by endothelial nitric oxide synthase (eNOS) located in the endothelial cell lining. Several chronic cardiovascular diseases such as hypertension, chronic kidney disease and diabetes are accompanied by endothelial dysfunction and hence diminished synthesis of NO. NO is a very reactive molecule and direct investigation of its function are limited and it has mainly been investigated by inhibition of eNOS. Recent research has shown that sodium nitrite is readily converted to NO by enzymes in vivo. The effects of sodium nitrite on renal variables, vasoactive hormones and central blood pressure are previously unexamined. It is now possible to achieve serial estimations of the central aortic systolic pressure (CASP) by a wrist born device.

Hypothesis:

1. Sodium nitrite infusion increases the urinary sodium excretion and glomerular filtration rate (GFR)
2. Sodium nitrite infusion increases plasma levels of nitrite, nitrate, NO and cyclic guanosine monophosphate (cGMP)
3. Sodium nitrite infusion lowers the peripheral and central blood pressure
4. Renal clearance of nitrite is constant and not dose dependent
5. Sodium nitrite infusion affects vasoactive hormones
6. The hemodynamic and renal effects is more pronounced in hypertensives as compared to healthy controls.

Purpose:

The purpose of this study is to investigate the effects of sodium nitrite infusion on

1. Renal handling of nitrite, nitrate, sodium and water
2. Plasma concentrations of vasoactive hormones
3. Peripheral (brachial) blood pressure and CASP

Design:

15 hypertensive subjects and 15 healthy, age and sex matched controls is recruited. Each subject will attend to two examination days. Four days prior to each examination day subjects are given a standardized diet with a low level of nitrate and nitrite. On the evening before the examination day the subjects take a single dose of lithium carbonate 300 mg in order to measure lithium clearance. On the examination days subjects are receiving a two hour infusion of either placebo (isotonic sodium chloride) or sodium nitrite. During the two examination days each subject receives both treatments in random order.

Perspectives:

Increasing knowledge about the nitrite-NO system can contribute to changing the clinical practise of diagnostics and treatment of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria (subjects with hypertension):

* BMI 18.5-30.0
* Ambulatory daytime blood pressure >135 mmHg systolic and/or >85 mmHg diastolic
* Women of childbearing potential must use safe contraception

Exclusion Criteria (subjects with hypertension):

* Tobacco smoking, medicine or substance abuse
* Weekly consumption of more than 14 units (12 g alcohol per unit) for women and 21 units for men
* Pregnancy or nursing
* Neoplasia
* Clinically significant heart, lung, liver, kidney, metabolic or neurologic disease
* Albuminuria > 300 mg/L
* Renography with signs of renal artery stenosis or hydronephrosis
* Clinically signs of secondary hypertension
* Clinically significant hypokalemia
* Clinically significant anemia
* Estimated glomerular filtration rate (eGFR) < 60 ml/min
* Clinically significant findings in screening blood samples, urine sample or ECG
* Persistent office blood pressure > 170/105 mmHg on the maximum dose of amlodipine (10 mg daily)
* Unacceptable symptoms of elevated blood pressure
* Unacceptable side effects of amlodipine

Inclusion Criteria (healthy normotensive subjects):

* BMI 18.5-30.0
* Women of childbearing potential must use safe contraception

Exclusion Criteria (healthy normotensive subjects):

* Tobacco smoking, medicine or substance abuse
* Weekly consumption of more than 14 units (12 g alcohol per unit) for women and 21 units for men
* Medical treatment 2 weeks prior to each examination day, except for contraception
* Pregnancy or nursing
* Neoplasia
* Clinically significant heart, lung, liver, kidney, metabolic or neurologic disease
* Clinically significant albuminuria
* Clinically significant anemia
* Estimated glomerular filtration rate (eGFR) < 60 ml/min
* Clinically significant findings in screening blood samples, urine sample or ECG
* Ambulatory daytime blood pressure >135/85 mmHg
* Blood donation within 1 month of the first examination day

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Fractional urinary sodium excretion (FENa) | 1 day

SECONDARY OUTCOMES:
Peripheral (brachial) blood pressure | 1 day
  Measured by oscillometric sphygmomanometer
Central aortic systolic blood pressure (CASP) | 1 day
  Measured by tonometric pulse wave analysis. Device BPro from HealthSTATS international, Singapore
Plasma concentration of nitrite and nitrate (NOx) | 1 day
Urinary excretion of nitrite and nitrate (NOx) | 1 day
Glomerular filtration rate | 1 day
Proximal sodium transport (Estimated by lithium clearance) | 1 day
  Estimated by lithium clearance
Free water clearance | 1 day
Urinary excretion of cyclic guanosine monophosphate (cGMP) | 1 day
Urinary excretion of epithelial sodium channels (ENaC) | 1 day
Urinary excretion of aquaporin 2 water channels (AQP2) | 1 day
Plasma concentration of renin (PRC) | 1 day
Plasma concentration of angiotensin II (ANG2) | 1 day
Plasma concentration of aldosterone | 1 day
Plasma concentration of atrial natriuretic peptide (ANP) | 1 day
Plasma concentration of brain natriuretic peptide (BNP) | 1 day
Plasma concentration of cyclic guanosine monophosphate (cGMP) | 1 day
Plasma concentration of endothelin | 1 day
Plasma concentration of vasopressin (AVP, ADH) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, MD, DMSc, Principal Investigator — Holstebro Regional Hospital
Locations (1):
- Department of Medical Research and Medicine, Holstebro Regional Hospital, Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Rosenbaek JB, Hornstrup BG, Jorgensen AN, Mortensen J, Pedersen EB, Bech JN. Effects of sodium nitrite on renal function and blood pressure in hypertensive vs. healthy study participants: a randomized, placebo-controlled, crossover study. J Hypertens. 2018 Mar;36(3):666-679. doi: 10.1097/HJH.0000000000001598. PMID 29065098